CLINICAL TRIAL: NCT02284581
Title: Evaluation of Medical Treatments (Chemotherapy, Hormonal Therapy and Biological Therapies) in Metastatic Breast Cancer Patients According to Biologic Subtype and Line of Treatment
Brief Title: Evaluation of Medical Treatments in MBC Patients According Biological Subtype and Line of Treatments
Acronym: BIO-META
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Consorzio Oncotech (Other)
Responsible Party: Sponsor
Other Study IDs: GIM14-BIOMETA
Record Dates: First submitted 2014-09-10; First posted 2014-11-06 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Breast Cancer
Keywords: MBC; metastatic; breast; observational; disease management
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: None Retained — Evaluation of duration of metastatic breast cancer treatments and numer of lines according to biological subtype (Luminal A, Luminal B, HER2 positive, triple-negative)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Retrospective cohort: All consecutive metastatic breast cancers patients treated in the participating site with a first-line therapy (chemotherapy or hormonal therapy with or without biological therapy) from last contact with patient or death which ever event comes first retrospectively back until 1st of January 2000.
- Prospective cohort: All new consecutive metastatic breast cancers patients will be treated in the participating site with a first-line therapy (chemotherapy or hormonal therapy with or without biological therapy) from site activation to June 2023.

SUMMARY:
Breast cancer is the most common cancer in many countries: in Italy about 48.000 new breast cancers are diagnosed every year and, despite improvements in diagnosis and therapy, about 13.000 women die every year for this disease . About 6-7% of breast cancer patients are metastatic at diagnosis , while the majority of patients with stage IV has a previous history of breast cancer that has already been treated. According to various prognostic factors (tumor size, lymph nodes involvement, grading, hormone receptors status, HER-2 status), in the worst-case scenario, more than 30% of node-negative breast cancer patients and more than 70% of node-positive patients relapse2.

The evolution of metastatic breast cancer has changed considerably in the last years with the approval of new drugs. In fact, already in 2003 Giordano et al showed that the prognosis of metastatic breast cancer patients was improved significantly from 1970's to 2000 with a median survival of 15 months in the early 1970's compared with 60 months in the last 1990's.

This significant survival gain was obtained with introduction of new drugs as hormonal, chemotherapeutic and biological agents. The greater availability of drugs has led to an increase in number of lines of treatment receiving by metastatic breast cancer patients. However, there are few published data on actual duration of metastatic breast cancer treatments. Moreover, there is no evidence to support a real impact on survival of treatments beyond the second-third line.

Recently, a retrospective analysis of about 199 metastatic breast cancer patients treated with chemotherapy showed that tumor subtype is associated with the duration and number of lines of chemotherapy (for example HER positive versus "triple-negative" patients) .

DETAILED DESCRIPTION:
The primary objectives are to evaluate the duration of metastatic breast cancer treatments (chemotherapy, hormonal therapy and biological therapies) according to biological subtype (Luminal A, Luminal B, HER2 positive, triple-negative) and to evaluate the number of lines of metastatic breast cancer treatments according to biological subtype (Luminal A, Luminal B, HER2 positive, triple-negative).

The secondary Objectives are to evaluate overall survival according to duration and to number of lines of metastatic breast cancer treatments and to identify predictive factors of number of lines of treatment as for example age, treatment response, biological subtype, metastatic sites, etc and to identify possible elements of different treatment management between participating sites.

The aim of this retrospective and prospective study is to identify the duration of treatments (chemotherapy, hormonal therapy and biological therapies) according to biological subtype and line of treatment in metastatic breast cancer patients.

An ancillary study will be conducted on part of population (HR+/HER2- patients newly diagnosed for mBC receiving first line CDk4/6 inhibitors).

For the ancillary study, it is expected to enroll at least 400 patients, who will be asked to fill in some questionnaires at the following visits, scheduled as per clinical practice:

* PROFFIT: baseline, day 1 cycle 3, day 1 cycle 5, every 6 months thereafter;
* Patient-reported outcomes (PRO): EORTC-QLQ-C30, FACT-B, COST-FACIT at baseline, day 1 cycle 3, day 1 cycle 5, every 6 months thereafter.

The ancillary study could evaluate:

* the impact of first line CDk4/6 inhibitors on HR+/HER2- metastatic breast cancer patients' financial toxicity
* retrospectively, the correlation between NLR and outcome in patients with breast cancer and in treatment with a CDk4/6 Inhibitor (as first line vs as second line)
* the correlation between BMI and outcome in patients with breast cancer and in treatment with a CDk4/6 Inhibitor (as first line vs as second line).

ELIGIBILITY:
Inclusion Criteria:

Retrospective cohort All consecutive metastatic breast cancers patients treated in the participating site with a first-line therapy (chemotherapy or hormonal therapy with or without biological therapy) from last contact with patient or death which ever event comes first retrospectively back until 1 st of January 2000

Prospective cohort All new consecutive metastatic breast cancers patients will be treated in the participating site with a first-line therapy (chemotherapy or hormonal therapy with or without biological therapy)from site activation to June 2023.

For the ancillary study

* Patients eligible for GIM 14 - BIO-META study
* HR+ HER2- patients newly diagnosed for mBC receiving CDk4/6 inhibitors as first-line or second-line treatment
* Written informed consent

Exclusion Criteria:

Not consecutive metastatic breast cancer patients grouped for a particular biological type (for example: all HER2 positive patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Italian patients with metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Duration and number of lines' treatment | Retrospectively from 2000 up to site activation; prospectively assested up to 32 months

SECONDARY OUTCOMES:
Overall Survival according duration | Retrospectively from 2000 up to site activation; prospectively assested up to 32 months
Overall survival according number of lines | Retrospectively from 2000 up to site activation; prospectively assested up to 32 months
Predictive factors of number of lines | Retrospectively from 2000 up to site activation; prospectively assested up to 32 months
Treatment management | Retrospectively from 2000 up to site activation; prospectively assested up to 32 months

OTHER OUTCOMES:
Impact of first line CDk4/6 inhibitors on HR+/HER2-mBC patients' financial toxicity | 30 months
Correlation between NLR and outcome in patients with breast cancer and in treatment with a CDk4/6 Inhibitor (as first line vs as second line) | 30 months
Correlation between BMI and outcome in patients with breast cancer and in treatment with a CDk4/6 Inhibitor (as first line vs as second line) | 30 months
Differences to the previously cited outcomes according to the type of CDk4/6 inhibitors | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Bighin, MD, Principal Investigator — IRCCS- Azienda Ospedaliera Universitaria San Martino-IST
Locations (35):
- Italy (35):
  - Centro di Riferimento Oncologico, Aviano
  - A.O. Consorziale Policlinico di Bari, Bari
  - A.O.U. Cagliari, Cagliari
  - Fondazione del Piemonte per l'Oncologia - I.R.C.C., Candiolo
  - Azienda Ospedaliera Ospedale Sant'Anna, Como
  - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - A.O.U. Sant'Anna, Ferrara
  - Ospedale 'F. Spaziani', Frosinone
  - Ospedale Policlinico San Martino IRCCS, Genova
  - A.O. Ospedale Civile di Legnano, Legnano
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST S.r.l., Meldola
  - ASST Fatebenefratelli Sacco - P.O. Fatebenefratelli, Milan
  - Ospedale Maggiore Policlinico - Fondazione IRCCS Ca' Granda, Milan
  - A.O.R.N. "A. Cardarelli", Napoli
  - Azienda ospedaliero universitaria "Federico II", Napoli
  - Istituto Nazionale per lo studio dei Tumori - Fondazione 'Pascale', Napoli
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Fondazione Maugeri IRCCS, Pavia
  - A.O.U. Pisana, Pisa
  - IRCCS Arcispedale Santa Maria Nuova, Reggio Emilia
  - Istituto Regina Elena per lo studio e la cura dei tumori, Roma
  - Policlinico Universitario A. Gemelli- DH Radiochemioterapia, Roma
  - Policlinico Universitario Agostino Gemelli, IRCSS-Unità Medicina di Precisione in Senologia, Roma
  - Policlinico Umberto I Università "La Sapienza" di Roma, Roma
  - Azienda Ospedaliera S. Andrea, Roma
  - Ospedale Sandro Pertini, Roma
  - Asl Roma 1 - Ospedale Santo Spirito, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera S. Andrea, Sassari
  - Ospedale Civile SS. Annunziata, Sassari
  - Ospedale 'SS. Trinità', Sora
  - A.O.U. Città della Salute e della Scienza di Torino - Presidio San Lazzaro, Torino
  - P.O. Martini - ASL TO1, Torino
  - ASL Alessandria - Ospedale Civile Santi Antonio e Margherita, Tortona
  - A.O.U. Santa Maria della Misericordia di Udine, Udine

REFERENCES:
- [Background] Cardoso F, Senkus-Konefka E, Fallowfield L, Costa A, Castiglione M; ESMO Guidelines Working Group. Locally recurrent or metastatic breast cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2010 May;21 Suppl 5:v15-9. doi: 10.1093/annonc/mdq160. No abstract available. PMID 20555067
- [Background] Schnipper LE, Smith TJ, Raghavan D, Blayney DW, Ganz PA, Mulvey TM, Wollins DS. American Society of Clinical Oncology identifies five key opportunities to improve care and reduce costs: the top five list for oncology. J Clin Oncol. 2012 May 10;30(14):1715-24. doi: 10.1200/JCO.2012.42.8375. Epub 2012 Apr 3. No abstract available. PMID 22493340
- [Background] Seah DS, Luis IV, Macrae E, Sohl J, Litsas G, Winer EP, Lin NU, Burstein HJ. Use and duration of chemotherapy in patients with metastatic breast cancer according to tumor subtype and line of therapy. J Natl Compr Canc Netw. 2014 Jan;12(1):71-80. doi: 10.6004/jnccn.2014.0008. PMID 24453294
- [Background] Goldhirsch A, Wood WC, Coates AS, Gelber RD, Thurlimann B, Senn HJ; Panel members. Strategies for subtypes--dealing with the diversity of breast cancer: highlights of the St. Gallen International Expert Consensus on the Primary Therapy of Early Breast Cancer 2011. Ann Oncol. 2011 Aug;22(8):1736-47. doi: 10.1093/annonc/mdr304. Epub 2011 Jun 27. PMID 21709140
- [Derived] Conte B, Fabi A, Poggio F, Blondeaux E, Dellepiane C, D'Alonzo A, Buono G, Arpino G, Magri V, Naso G, Presti D, Mura S, Fontana A, Cognetti F, Molinelli C, Pastorino S, Bighin C, Miglietta L, Boccardo F, Lambertini M, Del Mastro L; Gruppo Italiano Mammella (GIM) study group. T-DM1 Efficacy in Patients With HER2-positive Metastatic Breast Cancer Progressing After a Taxane Plus Pertuzumab and Trastuzumab: An Italian Multicenter Observational Study. Clin Breast Cancer. 2020 Apr;20(2):e181-e187. doi: 10.1016/j.clbc.2019.09.001. Epub 2019 Nov 14. PMID 31735691